CLINICAL TRIAL: NCT00856401
Title: Phase II Trial of Parathyroid Hormone for the Treatment of Hypoparathyroidism
Brief Title: ADD-ON Study to Existing Hypoparathyroidism Studies
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, John P Bilezikian, MD, MD, Columbia University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CFDA 93.103; NIH application ID 7566998 (Other Grant/Funding Number: FDA); CFDA 93.103 (Registry Identifier: CFDA 93103); FDA-002525-04A1 (Other: FDA - OOPD)
Record Dates: First submitted 2009-03-04; First posted 2009-03-05 (Estimated); Last update posted 2018-02-28 (Actual); Status verified 2018-02

CONDITIONS: Hypoparathyroidism
Keywords: hypoparathyroidism; hypopara; PTH; parathyroid hormone; CL-11-040; CL1-11 Study; NPSP 558; RELAY; RACE; REPLACE; HEXT; c10-007; c10-008; NPSP558; Columbia study; Columbia studies; HPTH; PTH1-84
MeSH Terms: conditions — Hypoparathyroidism | interventions — Parathyroid Hormone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- PTH1-84 in parent study (Experimental): In the RELAY, RACE, and HEXT study participants utilize PTH1-84. In the REPLACE Study participants utilize PTH1-84 or placebo of PTH1-84.
  Interventions: Drug: PTH1-84 in parent study

INTERVENTIONS:
Drug: PTH1-84 in parent study — daily injection of rhPTH(1-84); 25, 50 75, or 100mcg in parent study. In ADD-ON study, there is no intervention, only testing.
  Other Names: PTH1-84; PTH(1-84); rhPTH1-84; rhPTH(1-84); recombinant human parathyroid hormone 1-84

SUMMARY:
The purpose of this protocol is to add on additional exploratory studies to investigate changes in bone quality parameters with PTH(1-84) treatment of hypoparathyroidism. In addition to the biochemical hallmarks of hypoPT, it has been found that the microscopic structure of the bone, as well as the bone remodeling system, are markedly abnormal in this disease. How these abnormalities may be corrected with PTH(1-84) administration are not fully understood. The studies outlined in this add-on protocol are designed to shed light on the mechanistic ways that PTH(1-84) replacement may restore normal bone metabolism. These mechanistic studies are beyond the scope of the parent NPS study, which was designed to assess the safety and efficacy of PTH(1-84) in hypoPT treatment. Subjects who are participating in the NPS' REPLACE, RELAY, and RACE Studies and the HEXT Study at Columbia University will be invited to participate in this add-on protocol, which will involve a separate IRB-approved informed consent.

Study procedures:

1. High Resolution Peripheral Quantitative Computed Tomography (HRpQCT; XtremeCT, Scanco): Done at the same visit as DXA. In the REPLACE study twice, in RELAY once (or not at all if done within the last 6 months), in RACE twice, and in HEXT three times.
2. Osteolineage: At Baseline/Randomization/Visit One and at 4, 8, 12, 24, and 52 weeks of treatment in the REPLACE, RELAY, or RACE Study, if applicable, or at baseline and each 6-months visit in the HEXT Study, blood test for circulating osteogenic cells (10 cc) will be performed
3. Sclerostin: At Baseline/Randomization/Visit One and at 4, 8, 12, 24, and 52 weeks of treatment in the REPLACE, RELAY, or RACE Study, if applicable, or at baseline and each 6-months visit in the HEXT Study, blood test for sclerostin (5cc) will be performed

Funding Source - FDA OOPD

DETAILED DESCRIPTION:
In this protocol, we will investigate the mechanisms by which PTH(1-84) treatment improves bone quality in patients with hypoparathyroidism. Detailed imaging, cellular and biochemical studies will be performed on subjects with hypoparathyroidism who are also participating in the NPS Pharmaceutical Company's studies known as REPLACE, RELAY, RACE studies, and IND70449's HEXT Study. The parent NPS trial, being conducted under NPS's IND #76,514, is a multi-site, randomized, double-blind, placebo-controlled trial of PTH(1-84) in hypoparathyroidism. In the REPLACE Study, hypoparathyroid subjects are assigned to either placebo, 50, 75 or 100 mcg of PTH(1-84) a day, in a dose-titration design, for a 26 week period. In RELAY Study hypoparathyroid patients are randomized to 25mcg or 50mcg PTH1-84 for 8 weeks. In the RACE Study hypoparathyroid patients utilize 25, 50, 75, or 100mcg PTH1-84 for 52 weeks. The primary efficacy endpoint is a 50% reduction in calcium and calcitriol supplementation. The Columbia site is one of the investigative sites for the NPS protocol. A letter from NPS accompanying this document certifies that Dr. Bilezikian is a subinvestigator in the NPS project.

The protocol described in this proposal is different from the NPS study. It is being conducted under IND #70,449 to Dr. Bilezikian. It will pursue a number of additional studies that are not being sponsored by NPS or covered by their IND. Under IND #70,449 assigned to Dr. Bilezikian, we will investigate the effects of PTH(1-84) administration in hypoparathyroidism on bone quality in hypoparathyroidism. In addition to the biochemical hallmarks of hypoparathyroidism, it has been found that the microarchitectural structure of the bone and the entire bone remodeling system are markedly abnormal in this disease. The studies outlined in this add-on protocol are designed to elucidate the specific ways in which PTH(1-84) replacement restores to normal bone microstructure and bone metabolism in hypoparathyroidism. These mechanistic studies are beyond the scope of the parent NPS study, which is designed to assess only the safety and efficacy of PTH(1-84) in hypoparathyroidism. These special studies are being conducted only by Dr. Bilezikian's group at Columbia. In the summary which is provided here, we present the three major studies that will be conducted.

PROTOCOL #1: THE EFFECT OF PTH(1-84) ADMINISTRATION ON SKELETAL MICROSTRUCTURE AS DETERMINED BY HIGH RESOLUTION IMAGING OF THE SKELETON.[(PERIPHERAL QUANTITATIVE COMPUTED TOMOGRAPHY (HR-PQCT)).

Protocol. For all subjects enrolled at the Columbia site, we will perform HR-pQCT. Baseline measurement will be obtained twice at Visit 4 of the NPS protocol (2 weeks prior to randomization) and at Visit 16 of the NPS protocol (the final injection day). The reason for the duplicate measurements at each time point is to minimize any variance, thus improving the accuracy further of the data to be obtained.

Anticipated Results. Based upon our preliminary data, we expect that the abnormalities that we have observed at baseline in subjects with hypoparathyroidism will be improved by administration of PTH(1-84). The improvement in skeletal microstructure will be associated with greater bone strength as determined by finite element analysis and by individual assignment of strength to the specific orientation of trabecular plates and rods in the forearm and the tibia. In addition, the remarkable abnormalities in cortical structure will be a specific focus of attention, particularly in view of the fact that in a disease characterized by excessive secretion of PTH (primary hyperparathyroidism), cortical thinning is observed. Thus, with this add-on protocol, we will be able to test the hypothesis that PTH regulates the spatial distribution between cortical and trabecular bone. This anticipated result will add great value to the protocol and give us insights that would not otherwise be possible to make.

PROTOCOL #2: THE EFFECT OF PTH(1-84) ADMINISTRATION ON OSTEOBLAST CELLS AS DETERMINED BY MEASUREMENT OF CIRCULATING OSTEOGENIC PRECURSORS

Protocol. For all subjects enrolled in the NPS protocol at the Columbia site, we will perform measurements of peripheral circulating osteoblast cells. The assay will be performed at Visit 5 (randomization) of the NPS Protocol, then again at 4, 8, 12, and 24 weeks after administration of PTH(1-84).

Anticipated Results. Based upon our preliminary observations, we expect that PTH(1-84) will stimulate the recruitment, in the circulation, of cells with an osteoblastic phenotype. We expect that PTH(1-84) will also stimulate the maturation of cells as defined by ligand markers that can date the chronological age of these cells. The ability to demonstrate a specific osteoblastic effect on circulating cells will be correlated with changes in structural parameters to be obtained in these patients using HR-pQCT.

PROTOCOL #3: THE EFFECT OF PTH(1-84) ADMINISTRATION ON SCLEROSTIN, A KEY MEDIATOR OF PTH'S OSTEOANABOLIC ACTIONS.

Protocol. We will measure sclerostin levels at Visit 5 (randomization) of the NPS Protocol, then again at 4, 8, 12, and 24 weeks post-randomization. This will be the first time ever that sclerostin levels will be measured in hypoparathyroid subjects being replaced with PTH(1-84).

Anticipated Results. We expect that the administration of PTH(1-84) in subjects with hypoparathyroidism will be associated with acute reductions in sclerostin. By virtue of the experimental design of the study, we will be able to test further the kinetics of change, namely whether the anticipated acute fall in sclerostin levels will be sustained over time. The results can be related to the cellular actions of PTH to recruit and to activate the osteogenic cells that will be conducted in Protocol #2 as well as to the osteoanabolic effects we expect to demonstrate in Protocol #1. .

GENERAL STUDY FEATURES RELATED TO ALL PROTOCOLS

Enrollment and Eligibility Criteria. The enrollment criteria follow the protocol being sponsored by the NPS IND. They can be provided as an Appendix if requested. Study subjects who are enrolled in the NPS study will automatically be eligible for the protocols described above and will constitute the study population for these additional studies. We expect to enroll 16 patients for each of the remaining three years of the grant period.

Safety Measures. The safety measures to be conducted are identical to the NPS protocol sponsored under its IND #76,514. They can be provided as an Appendix if requested. They have been sent to the office of Dr. Mary Parks.

Overall Summary and Significance. These add-on protocols will be done uniquely at the Columbia site under the sponsorship of IND #70449 assigned to Dr. Bilezikian. They hold the promise of defining, in ways not possible by the standard protocol being sponsored by NPS, the mechanisms by which PTH(1-84) is therapeutic in subjects with hypoparathyroidism.

Funding Source - FDA OOPD

ELIGIBILITY:
Inclusion Criteria:

* active participation in the CL1-11-040, PAR-C10-007 or PAR-C10-008 Studies sponsored by NPS Pharmaceuticals.
* active participation in the HEXT Study of Dr. John Bilezikian.

Exclusion Criteria:

- not being a participant of the CL1-11-040, PAR-C10-007 or PAR-C10-008 Studies sponsored by NPS Pharmaceuticals or the HEXT Study of Dr. John Bilezikian.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2010-09; Primary Completion 2020-12-31 (Estimated); Study Completion 2021-06-30 (Estimated)

PRIMARY OUTCOMES:
HRpQCT | before and after treatment
  HPpQCT is performed twice in the REPLACE Study, one at Baseline, and again at 6 months. In the RELAY Study it is performed once at baseline, and only if it has not be done within the last 6 months. In the RACE study it is performed twice, once at baseline, then again at 52 weeks. In the HEXT study it is performed three times, once at baseline, then at 12 and 24 months.
sclerostin | variable depending on parent study
  At Baseline/Randomization/Visit One and at 4, 8, 12, 24, and 52 weeks of treatment in the REPLACE, RELAY, or RACE Study, if applicable, or at baseline and each 6-months visit in the HEXT Study. 5cc per draw.
circulating osteogenic precursors | variable depending on parent study
  At Baseline/Randomization/Visit One and at 4, 8, 12, 24, and 52 weeks of treatment in the REPLACE, RELAY, or RACE Study, if applicable, or at baseline and each 6-months visit in the HEXT Study. 10cc per draw.

CONTACTS AND LOCATIONS:
Overall Officials: John P Bilezikian, MD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Medical Center, New York, New York, United States